CLINICAL TRIAL: NCT03623906
Title: Comparison of Serrated Polyp Detection Rate Between Carbon Dioxide and Air Insufflation During Colonoscopy: a Randomized Controlled Multicenter Trial
Brief Title: Serrated Polyp Detection Rate Between Carbon Dioxide and Air Insufflation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, Dr, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SDR
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Serrated Polyp

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon dioxide insufflation colonoscopy (Experimental): Carbon dioxide insufflation colonoscopy
  Interventions: Procedure: Carbon dioxide insufflation colonoscopy
- Air insufflation colonoscopy (Active Comparator): Room air insufflation colonoscopy
  Interventions: Procedure: Air insufflation colonoscopy

INTERVENTIONS:
Procedure: Carbon dioxide insufflation colonoscopy — Carbon dioxide insufflation colonoscopy
  Arms: Carbon dioxide insufflation colonoscopy
Procedure: Air insufflation colonoscopy — Room air insufflation colonoscopy
  Arms: Air insufflation colonoscopy

SUMMARY:
Sessile serrated adenomas are characterized by their flat shape and the presence of a yellow mucus cap overlying the lesion. These morphological features may account for their diagnostic difficulty during colonoscopy. Missed proximal sessile serrated adenomas are regarded as an important cause for interval cancers in the right colon and emphasize the importance of developing quality measures intended to enhance their detection. There is only one single-center retrospective cohort study on the impact of carbon dioxide insufflation on the detection of serrated polyps during colonoscopy. The investigators designed a randomized, controlled trial to compare the effect of carbon dioxide insufflation vs. room air insufflation on serrated polyp detection rate.

ELIGIBILITY:
Inclusion Criteria:Patients 45-75-years-old who underwent a colonoscopy -

Exclusion Criteria:polyposis syndrome, Inflammatory bowel disease, previous colorectal operation

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Serrated polyp detection rate | 7 days